CLINICAL TRIAL: NCT02700633
Title: Does Permanent Pacemaker Status Confer Mortality Benefit in the Short Term Post TAVI
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Royal Sussex County Hospital (Other)
Responsible Party: Principal Investigator, David Hildick-Smith, Consultant Cardiologist, Royal Sussex County Hospital
Other Study IDs: TAVIPPMEarlyMortality
Record Dates: First submitted 2016-03-02; First posted 2016-03-07 (Estimated); Last update posted 2016-03-07 (Estimated); Status verified 2016-03

CONDITIONS: TAVI

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Those with pacemaker at discharge: Landmark analysis of early mortality dependant on pacemaker status at discharge
  Interventions: Device: Pacemaker
- Those without pacemaker at discharge: Landmark analysis of early mortality dependant on pacemaker status at discharge

INTERVENTIONS:
Device: Pacemaker
  Groups: Those with pacemaker at discharge

SUMMARY:
Pacemaker requirement in the immediate post procedure phase following TAVI is approximately 20% depending on device type and patient characteristics. There is a signal from recent studies suggesting increased risk of sudden cardiac / unexplained death in the first 30-60 days. This study aims to address whether there is a mortality advantage to having a pacemaker in the short term

ELIGIBILITY:
Inclusion Criteria:

* All patients post TAVI

Exclusion Criteria:

* Nil

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients post TAVI
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Actual)
Dates: Start 2016-02; Primary Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
30 day mortality | 30 dyas

SECONDARY OUTCOMES:
60 day mortality | 60 days